CLINICAL TRIAL: NCT00628147
Title: Tandem Colonoscopy Study of Narrow Band Imaging Versus White Light Examination to Compare Neoplasia Miss Rates
Brief Title: Clinical Evaluation of Narrow Band Imaging Colonoscope
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Roy Soetikno, Clinical Professor, VA Palo Alto Health Care System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: SOE0011
Record Dates: First submitted 2008-02-25; First posted 2008-03-04 (Estimated); Results first posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-01

CONDITIONS: Colonic Neoplasms
Keywords: colonic neoplasms; colonoscopy; narrow band imaging; diagnostic techniques
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Narrow band imaging colonoscope (Experimental): narrow band imaging colonoscope
  Interventions: Device: Narrow band imaging colonoscope
- White Light (No Intervention): Conventional White Light Examination

INTERVENTIONS:
Device: Narrow band imaging colonoscope — Adult colonoscopes with narrow band imaging capabilities (XCF-H160AY2L and XCF-Q160W6L, Olympus Medical Systems Corporation, Hachioji, Japan). There is an automatic switch on the handle of the endoscope that allows the physician to instantly switch between narrow band imaging and standard full spectrum white light modes.
  Other Names: CF-H180AL; CF-Q180AL; Evis Exera II CV-180
  Arms: Narrow band imaging colonoscope

SUMMARY:
The purpose of the study is to determine if colonoscopic examination using a colonoscope with a narrow band imaging light is more effective at detecting polyps compared to a colonoscope with standard full spectrum white light.

DETAILED DESCRIPTION:
This is a clinical study to evaluate whether the use of a new type of colonoscope may improve the detection of colon polyps. Though colonoscopy is currently the best test for colon cancer screening, it remains imperfect. Research has found that about 25% of polyps may actually be missed during colonoscopy using standard full spectrum white light imaging. Advances in colonoscopic technology hold the potential to decrease the miss rate of colorectal neoplasms. A new colonoscope uses narrow band imaging, whereby the colon is illuminated using only a subset of the white light spectrum, 415nanometers (blue) and 540 nanometers (green) rather than the standard full spectrum white light (red, green and blue). Initial studies by other groups suggest that these narrow band images highlight small blood vessels of colon polyps. As such, we hypothesized that the use of NBI would improve the identification of neoplasms through the color differentiation of precancerous or cancerous polyp (appearing brown) from normal colon mucosal lining (appearing green), and potentially lead to a reduction in polyp miss rate. We aimed to study the polyp miss rate, and compare narrow band imaging to white light examination.

ELIGIBILITY:
Inclusion Criteria:

* referred for elective outpatient colonoscopy

Exclusion Criteria:

* known inflammatory bowel disease
* personal or family history of polyposis syndrome
* referral for resection of a known lesion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2006-01; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Soetikno, MD, MS, Principal Investigator — VA Palo Alto Health Care System
Locations (1):
- VAPaloAltoHCS, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kaltenbach T, Friedland S, Soetikno R. A randomised tandem colonoscopy trial of narrow band imaging versus white light examination to compare neoplasia miss rates. Gut. 2008 Oct;57(10):1406-12. doi: 10.1136/gut.2007.137984. Epub 2008 Jun 3. PMID 18523025

RESULTS

PARTICIPANT FLOW:
Groups:
- Narrow Band Imaging Colonoscope: Narrow band imaging colonoscope (CF-H180AL, CF-Q180AL, Evis Exera II CV-180): Adult colonoscopes with narrow band imaging capabilities (XCF-H160AY2L and XCF-Q160W6L, Olympus Medical Systems Corporation, Hachioji, Japan). There is an automatic switch on the handle of the endoscope that allows the physician to instantly switch between narrow band imaging and standard full spectrum white light modes.
Period: Overall Study
Arm/Group | Narrow Band Imaging Colonoscope | White Light
Started | 142 | 142
Completed | 135 | 141
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Narrow Band Imaging Colonoscope | White Light | Total
Number analyzed (Participants) | 142 | 142 | 284
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10) | 64 (10) | 64 (10)
Gender [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 137 | 138 | 275

OUTCOME MEASURES:

1. Primary Outcome: Neoplasm Miss Rate
Time Frame: same day
Measure: Number (95% Confidence Interval); unit: Miss rate percentage
Arm/Group | Narrow Band Imaging Colonoscope | White Light
Number analyzed (Participants) | 135 | 141
Miss rate percentage | 12.6 [7.5 to 19.4] | 12.1 [7.2 to 18.6]

2. Secondary Outcome: Neoplasm Detection Rates
Time Frame: same day
Population: We report overall neoplasia detection rate, and then report a sub-analysis for the neoplasia detection rates by indication (screening vs non-screening).
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Band Imaging Colonoscope | White Light
Number analyzed (Participants) | 135 | 141
Participants
  Overall | 69 | 66
  Screening: number analyzed (Participants) | 66 | 67
  Screening | 29 | 31
  Non-Screening: number analyzed (Participants) | 69 | 74
  Non-Screening | 40 | 35

3. Secondary Outcome: Completion of Examinations
Time Frame: same day
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Band Imaging Colonoscope | White Light
Number analyzed (Participants) | 135 | 141
Participants | 135 | 141

4. Secondary Outcome: Procedure Complications
Time Frame: procedure and post-procedure complications within 30 days after colonoscopy
Measure: Count of Participants; unit: Participants
Arm/Group | Narrow Band Imaging Colonoscope | White Light
Number analyzed (Participants) | 135 | 141
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Narrow Band Imaging Colonoscope | White Light
Serious Adverse Events (participants affected / at risk) | 0/142 | 0/142
Other Adverse Events (participants affected / at risk) | 0/142 | 0/142

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No